CLINICAL TRIAL: NCT04892238
Title: Helicobacter Pylori Infection Occurrence in Primary Care Settings in Russia
Brief Title: Helicobacter Pylori Infection Occurrence in Russia
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Collaborators: Moscow Clinical Scientific Center (Other); St. Petersburg State Pavlov Medical University (Other); People's Friendship University of Russia (Other)
Responsible Party: Principal Investigator, Sergey Morozov, Leading researcher, Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Other Study IDs: АААА-А18-118021590202-9; АААА-А18-118021590202-9 (Registry Identifier: NIOKTR ROSRID); АААА-А17-117080910167-9 (Registry Identifier: NIOKTR ROSRID)
Record Dates: First submitted 2021-05-13; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; occurrence; ambulatory settings; prospective trial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment-naïve: Subjects without previous experience of treatment provided for H.pylori infection
  Interventions: Diagnostic Test: 13-C urea breath test
- treatment experienced: Subjects who were previously tested positive for H.pylori infection and who were treated for H.pylori infection with at least 2 antibiotics in combination with proton pump inhibitor not less than 6 weeks before the 13C-urea breath test
  Interventions: Diagnostic Test: 13-C urea breath test

INTERVENTIONS:
Diagnostic Test: 13-C urea breath test — Standard urea breath test (UBT) ("HELICARB", LLC "ISOCARB", reg. cert. #РЗН 2016/3773 issued by Roszdravnadzor on 29.02.2016) with 13C-carbamide of 99% purity used for the study.
  Samples of exhaled air obtained before and after 20 minutes after 50 mg 13C-urea intake are analysed for 13C/12C isotope ratio with the use of infrared spectrometer "IRIS.Doc" (Kibion, Sweden). Delta over baseline (δ) of 13C / 12C is calculated based on the results of the initial and second samples, the results were shown in ppm (‰). The results of the test is negative if δ was <4.0‰; test results with δ ≥4.0‰ are considered positive.

SUMMARY:
This study is planned to reveal the occurrence rate of H.pylori infection in ambulatory settings' patients in Russia and to compare the occurrence rates in different years in treatment-naïve and previously treated subjects.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate (based on the signed informed consent form);
* age older than 12 y.o. (for subjects younger than 18 y.o. written informed consent of a legal representative was obligatory);
* availability of demographic data and medical history, including previous treatment for H.pylori infection

For subjects of "treatment-naïve" group:

* no previous treatment for H.pylori infection in the anamnesis;
* at least 6 weeks after previous use of any antimicrobial agents for any reason;
* at least 2 weeks' time frame free of use of proton pump inhibitors, other anti-secretory agents and bismuth preparations.

For "Previously treated" group of subjects:

* infection caused by H.pylori established earlier and
* not less than 6 weeks after the end of eradication therapy with at least 2 antibiotics and a proton pump inhibitor for at least 7 days, based on a patient's report

Exclusion Criteria:

* history of surgery on chest, stomach, gut (excluding appendectomy or laparoscopic cholecystectomy performed more than 6 month before the enrolment);
* advanced stage of chronic obstructive pulmonary disease,
* allergies to citruses,
* pregnant and breastfeeding women.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Ambulatory subjects, referred to perform urea breath test (UBT) and who gave written informed consent for the use of their data for research purposes are aligible for the study.
Sampling Method: Probability Sample
Enrollment: 70000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Presence of H.pylori infection | during the procedure
  Delta over the baseline (δ) of 13C/12C based on the results of the initial and second samples ≥4.0‰ are positive

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Bordin, MD, PhD, Professor, Principal Investigator — Moscow Clinical Scientific Center
Locations (2):
- Russia (2):
  - Moscow Clinical Scientific Center, Moscow
  - Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology, Moscow

IPD SHARING:
Plan to Share IPD: Yes
Depersonalised data will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon request
Access Criteria: reasonable request to the principal investigator
URL: http://ion.ru

REFERENCES:
- [Derived] Bordin D, Morozov S, Plavnik R, Bakulina N, Voynovan I, Skibo I, Isakov V, Bakulin I, Andreev D, Maev I. Helicobacter pylori infection prevalence in ambulatory settings in 2017-2019 in RUSSIA: The data of real-world national multicenter trial. Helicobacter. 2022 Oct;27(5):e12924. doi: 10.1111/hel.12924. Epub 2022 Aug 16. PMID 35971900